CLINICAL TRIAL: NCT01424878
Title: Study of Molecular Pathways in Medullary Thyroid Carcinoma (MTC) and Correlation of Molecular Data With Clinical Behavior of the MTC in Individuals Patients
Brief Title: Study of Molecular Pathways in Medullary Thyroid Carcinoma and Correlation of Molecular Data With Clinical Behavior of the MTC in Individuals Patients
Status: Completed | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999910167; 10-C-N167
Record Dates: First submitted 2011-08-26; First posted 2011-08-29 (Estimated); Last update posted 2018-04-05 (Actual); Status verified 2014-02-12

CONDITIONS: Medullary Thyroid Carcinoma; Multiple Endocrine Neoplasia Type 2
Keywords: Molecular Analysis of Medullary Thyroid Carcinoma Tissues
MeSH Terms: conditions — Carcinoma, Medullary; Multiple Endocrine Neoplasia Type 2a

STUDY DESIGN:
Time Perspective: Retrospective

SUMMARY:
Background:

Medullary thyroid carcinoma (MTC) is a rare malignancy, occurring either as a sporadic disease (75% of cases), or in a hereditary pattern as multiple endocrine neoplasia (MEN) type 2 (MEN2A or MEN2B) or familial medullary thyroid carcinoma (FMTC). The MTC arises from the neural crest C-cells and in hereditary cases the first pathological disorder is C-cell hyperplasia (CCH) Most patients with MTC have advanced disease at the time of diagnosis.

Chemotherapy and external beam radiotherapy have been minimally effective. Molecular targeted therapeutics (MTTs) and other receptor kinases in patients with advanced MTC have demonstrated activity.

Despite some clinical responses, the collection of tumor tissues and autologous normal tissues has been virtually non-existent. Thus, laboratory studies defining affected molecular targets and downstream pathways, and molecular data providing direction for future clinical trials has yet to occur.

Data from molecular studies of tumor tissue of hereditary or sporadic MTC patients will assist in predicting clinical behavior and the biology of MTC in predicting response to a given MTT, and in designing combination clinical trials.

Objectives:

Clarify how normal molecular pathways are altered by mutations in the RET protooncogene. Including additional genetic mutations and unidentified chromosomal translocations.

Correlate results from molecular analyses of MTC tissue with patient s clinical course.

Define how the molecular and clinical data will be useful in designing targeted therapy for patients with MTC.

Eligibility:

Patients must have confirmed diagnosis of C-cell hyperplasia, primary MTC, or metastatic MTC with archived pathology specimens available at Washington University.

Design:

Paraffin blocks of MTC tissues from archival samples at Washington University Department of Pathology will be selected.

H&E slide from selected tissue blocks will be examined for molecular study suitability.

Necessary tissue samples from blocks will have molecular studies, including, gene arrays, array comparative genomic hybridization, immunohistochemistry, and sequencing.

Retrospective chart review will occur to obtain relevant clinical information.

DETAILED DESCRIPTION:
Background:

Medullary thyroid carcinoma (MTC) is a rare malignancy, occurring either as a sporadic disease (75% of cases), or in a hereditary pattern as multiple endocrine neoplasia (MEN) type 2 (MEN2A or MEN2B) or familial medullary thyroid carcinoma (FMTC). The MTC arises from the neural crest C-cells and in hereditary cases the first pathological disorder is C-cell hyperplasia (CCH) Most patients with MTC have advanced disease at the time of diagnosis.

Chemotherapy and external beam radiotherapy have been minimally effective. Molecular targeted therapeutics (MTTs) and other receptor kinases in patients with advanced MTC have demonstrated activity.

Despite some clinical responses, the collection of tumor tissues and autologous normal tissues has been virtually non-existent. Thus, laboratory studies defining affected molecular targets and downstream pathways, and molecular data providing direction for future clinical trials has yet to occur.

Data from molecular studies of tumor tissue of hereditary or sporadic MTC patients will assist in predicting clinical behavior and the biology of MTC in predicting response to a given MTT, and in designing combination clinical trials.

Objectives:

Clarify how normal molecular pathways are altered by mutations in the RET protooncogene. Including additional genetic mutations and unidentified chromosomal translocations.

Correlate results from molecular analyses of MTC tissue with patient s clinical course.

Define how the molecular and clinical data will be useful in designing targeted therapy for patients with MTC.

Eligibility:

Patients must have confirmed diagnosis of C-cell hyperplasia, primary MTC, or metastatic MTC with archived pathology specimens available at Washington University.

Design:

Paraffin blocks of MTC tissues from archival samples at Washington University Department of Pathology will be selected.

H&E slide from selected tissue blocks will be examined for molecular study suitability.

Necessary tissue samples from blocks will have molecular studies, including, gene arrays, array comparative genomic hybridization, immunohistochemistry, and sequencing.

Retrospective chart review will occur to obtain relevant clinical information.

ELIGIBILITY:
* INCLUSION CRITERIA:

Patients must have confirmed diagnosis of C-cell hyperplasia, primary MTC, or metastatic MTC with archived pathology specimens available at Washington University.

Ages: 2 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2010-07-05; Study Completion 2014-02-12

CONTACTS AND LOCATIONS:
Overall Officials: Antonio T Fojo, M.D., Principal Investigator
Locations (1):
- National Cancer Institute (NCI), 9000 Rockville Pike, Bethesda, Maryland, United States